CLINICAL TRIAL: NCT00253890
Title: Insomnia and Drug Relapse Risk
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael Stein, MD, Director, General Medicine Research, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01DA020479 (NIH); R01DA020479-01 (NIH)
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-10

CONDITIONS: Poor Quality Sleep; Opiate Addiction
Keywords: sleep quality; methadone; substance use
MeSH Terms: conditions — Opioid-Related Disorders; Sleep Initiation and Maintenance Disorders; Substance-Related Disorders | interventions — Trazodone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trazodone (Active Comparator): 50-150mg (50mg capsules) at bedtime for 90 days
  Interventions: Drug: Trazodone
- Placebo (Placebo Comparator): 1-3 capsules at bedtime for 90 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trazodone — 50 mg 1-3 capsules at bedtime for 3 months
  Other Names: Desyrel; Oleptro; Beneficat; Deprax; Desirel; Molipaxin; Thombran; Trazorel; Trialodine; Trittico; Mesyrel
  Arms: Trazodone
Drug: Placebo — 1-3 at bedtime
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purposes of this study are:

1. to evaluate the relationship between subjective complaints of sleep and objective measures of sleep quality, as measured through polysomnography, and
2. to evaluate the efficacy of trazodone, as compared to placebo, in individuals early in methadone maintenance.

DETAILED DESCRIPTION:
Individuals new to methadone maintenance will be asked to participate in this 6-month, double-blind, randomized control trial. All participants will complete a baseline interview, a medical screening and follow-up interviews at 1, 3 and 6-months post-baseline. These interviews take approximately 60 minutes, and survey various areas of the participants' experiences, including basic demographic information, mood, sleep and substance use areas. All participants will also be asked to complete a 2-night sleep monitoring at the time of the baseline interview and again at the 1-month follow-up interview. Participants will also receive study medication; half of the participants will receive a placebo medication, and the other half will receive Trazodone, a widely-prescribed, well-tolerated, low side-effect medication. Neither the participant nor the study staff will know which medication the participant is taking while the participant is actively enrolled in the study. This information can be available to the participant at the end of his/her study participation.

ELIGIBILITY:
Inclusion Criteria:

* Recent methadone maintenance enrollment
* Sleep complaints as measured by the Pittsburgh Sleep Quality Index (PSQI)
* No medical contraindications to trazodone

Exclusion Criteria:

* Methadone maintenance enrollment not recent
* No sleep complaints as measured by the PSQI
* Medical contraindications to trazodone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2005-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Stein, MD, Principal Investigator — Rhode Island Hospital; Rogers Griffith, MD, Study Director — The Miriam Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Kurth ME, Sharkey KM, Millman RP, Corso RP, Stein MD. Insomnia among methadone-maintained individuals: the feasibility of collecting home polysomnographic recordings. J Addict Dis. 2009 Jul;28(3):219-25. doi: 10.1080/10550880903014155. PMID 20155590

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 8 methadone maintenance clinics in the Providence, RI area.
Groups:
- Trazodone: 50-150mg at bedtime
- Placebo: 1-3 capsules at bedtime
Period: Overall Study
Arm/Group | Trazodone | Placebo
Started | 69 | 68
Completed | 62 | 61
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trazodone | Placebo | Total
Number analyzed (Participants) | 69 | 68 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 69 | 68 | 137
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.0 (8.8) | 38.5 (8.7) | 38.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 39 | 73
  Male | 35 | 29 | 64
Region of Enrollment [Number; unit: participants]
  United States | 69 | 68 | 137

OUTCOME MEASURES:

1. Primary Outcome: Sleep Quality, as Measured by Total Sleep Time
Description: Number of minutes spent sleeping during sleep period, as measured by daily sleep diary.
Time Frame: Baseline to 1-month
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Trazodone | Placebo
Number analyzed (Participants) | 67 | 67
minutes | 339 (136) | 329 (124)
Statistical Analysis 1: Comparison: Trazodone vs Placebo; Change in sleep quality was assessed by calculating gain scores. We used a 2-sided t-test to report mean change; Test type: Superiority or Other; p = .05, t-test, 2 sided; Mean Difference (Net) = 35.7

ADVERSE EVENTS:
Arm/Group | Trazodone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/68
Other Adverse Events (participants affected / at risk) | 0/69 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No